CLINICAL TRIAL: NCT03149367
Title: Fixed Versus Adjustable Sutures in Management of Blepheroptosis
Brief Title: Surgical Management of Blepharoptosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Ali Essameldeen Mohamed Ali, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7540
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Blepharoptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed suture (Experimental)
  Interventions: Procedure: levator muscle resection with fixed sutures technique
- Adjustable suture (Experimental)
  Interventions: Procedure: Levator muscle resection with adjustable sutures technique

INTERVENTIONS:
Procedure: levator muscle resection with fixed sutures technique — The levator muscle is approached through skin incision and the muscle shortened and sutured directly to the tarsus then the skin crease reformed with interrupted sutures which pick up the underlying levator muscle
  Arms: Fixed suture
Procedure: Levator muscle resection with adjustable sutures technique — The adjustable sutures technique in which the sutures passes through the levator muscle into the tarsal plate and out through the skin edge .the skin crease is formed separately so that adjusting the suture doesn't open the wound, the suture can be adjusted according to the result up to 4 days post operative.
  Arms: Adjustable suture

SUMMARY:
Comparison of the results of levator resection operation with the use of fixed sutures technique in which the levator muscle is approached through skin incision and the muscle shortened and sutured directly to the tarsus then the skin crease reformed with interrupted sutures which pick up the underlying levator muscle versus the results with the use of adjustable sutures in which the suture passes through the levator muscle into the tarsal plate and out through the skin edge .the skin crease is formed separately so that adjusting the suture doesn't open the wound, the suture can be adjusted according to the result up to 4 days post operative.

ELIGIBILITY:
Inclusion criteria:

* Cases of blepharoptosis admitted at Assiut University Hospital.
* Cases that are fit for surgery.

Exclusion criteria:

* Cases not fit for surgery.
* Cases of pseudoptosis may result from many conditions that simulate an asymmetry of the upper eyelid level. Dysthyroid ophthalmopathy, enophthalmos, or exophthalmos can accentuate a minimal blepharoptosis or produce the appearance of blepharoptosis on the contralateral normal side,
* Cases with diseases, such as myasthenia gravis; negativity for Bell palsy symptoms; and Marcus Gunn jaw-winking syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
The cosmetic appearance | One week
  Symmetry of the two eyelids was calculated based on the difference in the margin reflex distance between them in the primary position of gaze. The results were classified into good, fair, and poor

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university hospital, Asyut, Egypt